CLINICAL TRIAL: NCT06116214
Title: Effect of Vachellia Nilotica Versus Sodium Hypochlorite as Root Canal Irrigant on Postoperative Pain and Bacterial Load Reduction in Mandibular Premolar Teeth With Necrotic Pulp
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gozlan Fouad Saad Mohamed, Principal Investigator, master's degree student, Endodontic Department, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFSMohamed
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Necrotic Pulp; Post Operative Pain
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): in this group the teeth will be irrigated with 2.5% Sodium Hypochlorite (gold standard)
  Interventions: Other: sodium hypochlorite
- Experimental group (Experimental): in this group the teeth will be irrigated with 10% V. Nelotica (Herbal irrigant)
  Interventions: Other: Vachellia Nelotica

INTERVENTIONS:
Other: Vachellia Nelotica — As a root canal irrigant (herbal)
  Other Names: Babul
  Arms: Experimental group
Other: sodium hypochlorite — As a root canal irrigant
  Arms: Control group

SUMMARY:
The aim of this study is to assess the effect of V. nilotica extract solution versus 2.5% NaOCl on the intensity of postoperative pain and the amount of bacterial load reduction.

DETAILED DESCRIPTION:
Clinical compare the effect of V. nilotica extract solution versus 2.5% NaOCl on the intensity of postoperative pain and the amount of bacterial load reduction when used as root canal irrigant in necrotic pulp. The post operative pain will be recorded using Numerical rating scale, and the bacterial load reduction will be measured by Bacterial counting using agar culture technique.

ELIGIBILITY:
Inclusion criteria:

1. Systemically healthy patient (ASA I, II).
2. Age between 20 and 40 years.
3. Male or female.
4. Patient who is able to sign and comprehend the pain scale (committed patient).
5. Mandibular single rooted premolars having the following criteria:

   * With single root canal.
   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pulpal pain.
   * Positive pain on percussion denoting apical periodontitis.
   * Slight widening of periodontal space or peri-apical radiolucency smaller than 3 mm (0-2mm).

Exclusion criteria:

1. Medically compromised patients (ASA III or IV).
2. Teeth with:

   * Immature roots.
   * Vital pulp tissues.
   * Association with swelling.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III.
   * Previously accessed or endodontically treated.
   * Deep periodontal pockets more than 4 mm.
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
3. Patients who could not interpret the NRS.
4. Patients with diabetes, immune-compromising, and immunosuppression disease and pregnant women will be also excluded.
5. History of intolerance to NSAIDs.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
post operative pain. | At 6, 12, 24, and 48 hours postoperatively (post instrumentation and post obturation)
  non=0, mild=1-3, moderate4-6, sever=7-10. Measured and reported by Numerical Rating Scale (NRS). Minimum value=0, maximum value=10, the higher score or value mean a worse outcome.

SECONDARY OUTCOMES:
Bacterial load reduction | 1 hour. First sample (S1) will be taken pre-intervention (before chemo-mechanical preparation) and the second sample (S2) will be taken immediately after the intervention (after completion of chemo-mechanical preparation) on the same visit.
  Bacterial counting using agar culture technique.

CONTACTS AND LOCATIONS:
Overall Officials: Gozlan FS Mohamed, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No
Not chosen yet